CLINICAL TRIAL: NCT07049510
Title: The Effect of the Programme on Combating Violence Against Women on Domestic Violence Awareness and Gender Attitudes: A Randomized Controlled Trial
Brief Title: Combating Violence Against Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, PhD, Hitit University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: Combating Violence Against Wom
Record Dates: First submitted 2025-06-13; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Nursing Role

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: Control group (Active Comparator): All women will be given the Personal Information Form, Domestic Violence Awareness Scale and Gender Role Attitude Scale as a pre-test. No intervention will be made to the control group. After 8 weeks, all women will be reunited and given the Domestic Violence Awareness Scale and Gender Role Attitude Scale as a post-test.
  Interventions: Behavioral: Experimental: Experimental: Combating violence against women
- Combating violence against women (Experimental): After the Personal Information Form, Domestic Violence Awareness Scale and Gender Role Attitude Scale are applied to all women as a pre-test, the women in the experimental group will be included in the Combating Violence Against Women program. The program will be given in 4 sessions in 1 day. Demonstration, powerpoint, feedback and brainstorming methods will be used in the training.
  8 weeks after the completion of the training, all women will be reunited and the Domestic Violence Awareness Scale and Gender Role Attitude Scale will be applied as a post-test.
  Interventions: Behavioral: Experimental: Experimental: Combating violence against women

INTERVENTIONS:
Behavioral: Experimental: Experimental: Combating violence against women — After the Personal Information Form, Domestic Violence Awareness Scale and Gender Role Attitude Scale are applied to all women as a pre-test, the women in the experimental group will be included in the Combating Violence Against Women program. The program will be given in 4 sessions in 1 day. Demonstration, powerpoint, feedback and brainstorming methods will be used in the training.
  8 weeks after the completion of the training, all women will be reunited and the Domestic Violence Awareness Scale and Gender Role Attitude Scale will be applied as a post-test.

SUMMARY:
The aim of the study was to investigate the effect of the program to combat violence against women on domestic violence awareness and gender role attitudes.

DETAILED DESCRIPTION:
Personal Information Form, Domestic Violence Awareness Scale and Gender Role Attitude Scale will be used in collecting research data.

After the Personal Information Form, Domestic Violence Awareness Scale and Gender Role Attitude Scale are applied to all women as a pre-test, the women in the experimental group will be included in the Combating Violence Against Women program. The program will be given in 4 sessions in 1 day. Demonstration, powerpoint, feedback and brainstorming methods will be used in the training.

No intervention will be made to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-45,
* Who speaks Turkish,
* Who has previously applied to law enforcement due to violence,
* Women who volunteer to participate in the research.

Exclusion Criteria:

* Women diagnosed with a psychiatric illness.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Domestic Violence Awareness Scale | 2 months
  The scale developed by Özyürek and Kurnaz (2019) consists of 20 items measuring awareness of domestic violence on a three-point Likert scale. The highest score that can be obtained from each item is three, and the lowest score is one. Items 1-5 in the scale constitute the sub-dimensions of "Definition of Domestic Violence", items 6-10 constitute the sub-dimensions of "Consequences of Domestic Violence", items 11-15 constitute the sub-dimensions of "Acceptance of Domestic Violence", and items 16-20 constitute the sub-dimensions of "Normalization of Domestic Violence". High total scores obtained from the entire scale can be interpreted as the individual having views compatible with the expected behaviors and attitudes in scientific and legal fields in interpreting domestic violence and having a high level of awareness of domestic violence. The Cronbach alpha coefficient of the scale was reported to be 0.92 and ranged between 0.71 and 0.92 for its sub-dimensions. In this study, Cronbach

SECONDARY OUTCOMES:
Gender Roles Attitude Scale | 2 months
  Gender Roles Scale was originally developed by García-Cueto and colleagues (2015). Adaptation of the scale to Turkish and reliability validity study were conducted by Bakioğlu and Türküm (2019). In the original study, Cronbach alpha internal consistency coefficient was calculated as 0.99 within the scope of reliability of the scale, in the adaptation study, Cronbach alpha internal consistency coefficient was calculated as 0.88 and test-retest reliability was calculated as 0.77. The scale consists of 15 questions and a single dimension. The items are answered in Likert type as 1= I completely disagree, 2= I disagree, 3= I am undecided, 4= I agree, 5= I completely agree and so on. The 13 items of the scale, except for items 1 and 2, are reverse coded. A total score is obtained from the scale, and a higher score indicates a higher negative attitude towards gender roles. In other words, a person who scores high on the scale adopts gender roles less and shows less commitment than a person

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared with researchers who apply for appropriate use for research purposes only, with ethics committee approval.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after publication
Access Criteria: Researchers who are conducting research in the same field and have received ethics committee approval.
URL: http://Currently_not_available.